CLINICAL TRIAL: NCT02489331
Title: Post Marketing Surveillance of Safety and Efficacy for Cholib® in Korean Patients Under the "New Drug Re-examination".
Brief Title: Post Marketing Surveillance of Safety and Efficacy for Cholib in Korean Patients Under the "New Drug Re-examination".
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: FESI5001
Record Dates: First submitted 2015-06-24; First posted 2015-07-03 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Dyslipidemias
Keywords: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Post marketing surveillance of safety and efficacy for Cholib in Korean patients under the "New Drug Re-examination"

DETAILED DESCRIPTION:
The objective of this surveillance is to identify problems and questions on Cholib® and on the following matters under the condition that the investigational product is in use.

1. Serious adverse event and adverse drug reaction profile

   * Death or a life-threatening condition
   * Hospitalization or prolonged hospitalization
   * Persistent or significant disability/incapacity
   * Congenital anomaly/birth defect
   * Other medically significant events
2. Unexpected adverse event/adverse drug reaction profile
3. Known adverse drug reaction profile
4. Non-serious adverse drug reaction profile
5. Other information related to the product safety
6. Efficacy evaluation
7. Study of extended follow-up Surveillance of the safety and efficacy of the subjects who received Cholib® for long-term use at least 24 weeks.
8. Study of special patient Analysis of specific patients such as elderly patients (65 years and above), patients with renal/hepatic disease

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of mixed dyslipidaemia who has high triglycerides and low HDL cholesterol level while LDL cholesterol levels are adequately controlled with the corresponding dose of simvastatin monotherapy

Exclusion Criteria:

* Patients who are hypersensitive (allergic) to peanuts, soybean or any of the ingredients of the medicine
* Patients who experienced photoallergy or phototoxic reactions during treatment with fibrates or ketoprofen
* Patients who have active hepatic disorder or have serum transaminase increased continuously without identified reason
* Patients who have gallbladder disease
* Patients who have chronic or acute pancreatitis except acute pancreatitis due to severe hypertriglyceridemia
* Patients who have moderately or severely reduced kidney function(estimated glomerular filtration rate < 60mL/min/1.73m2)
* Cholib® administration combined administration with fibrates, statins, danazol, cyclosporine or strong cytochrome P450(CYP)3A4 inhibitor
* 145/40mg Cholib® Combined administration with amiodarone, verapamil, amlodipine or diltiazem
* Children <19 years
* Pregnant or breast-feeding women
* Patients with biliary cirrhosis
* Patients who have myopathy and/or previously had rhabdomyolysis or myopathy while taking statins and/or fibrates or had 5 times more creatine phosphokinase than Upper limit of Normal (ULN) while taking statins previously
* Patients who have rare hereditary problems with lactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption since this drug contains lactose
* Patients who have rare hereditary problems with fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase deficiency since this drug contains sucrose
* Patients who have LDL Cholesterol ≥130 mg/dL and triglyceride < 150mg/dL and HDL cholesterol ≥60mg/dL Investigators will refer to the product market authorization (label) for inclusion/exclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are prescribed Cholib as per doctor's medical judgement in normal medical parctice setting
Sampling Method: Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse event after Cholib administration in general medical practice | 24 weeks
  Any adverse events occurred after Cholib® dosing will be recorded. Description of adverse event(s) including type of adverse event(s), onset/end date, severity, action taken, causal relationship to the drug and investigator's view on the adverse event(s) will be captured, whether it is related to the drug or not and until follow up visit more than 1 time during the surveillance period.
  Lab abnormalities and changes in vital signs are considered to be adverse events only if they result in discontinuation from the study, necessitate therapeutic medical intervention, and/or if the investigator considers them to be adverse events.
Incidence of serious adverse event after Cholib administration in general medical practice | 24 weeks
  Any serious adverse events occurred after Cholib® dosing will be recorded. Description of serious adverse event(s) including type of serious adverse event(s), onset/end date, severity, action taken, causal relationship to the drug and investigator's view on the serious adverse event(s) will be captured, whether it is related to the drug or not and until follow up visit more than 1 time during the surveillance period.
  Lab abnormalities and changes in vital signs are considered to be serious adverse events only if they result in discontinuation from the study, necessitate therapeutic medical intervention, and/or if the investigator considers them to be serious adverse events.

SECONDARY OUTCOMES:
Evaluate four categories based on Serum-Triglyceride, HDL cholesterol, LDL cholesterol, creatine kinase (CK), alanine aminotransferase (ALT), aspartate aminotransferase (AST) and creatinine level after Cholib® dosing and test date | 24 weeks
  All subjects who received Cholib® for at least 12 weeks and follow-up at 24 weeks will be evaluated for efficacy using the four-criteria as follows:
  Improved, unchanged, exacerbated, not assessable

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Daesung Medical Center, Bucheon-si
  - Isam Clinic, Busan
  - DongRae BongSeng Hospital, Busan
  - Hyundai Medical Clinic, Daegu
  - SANGIN Clinic of Internal Medicine, Daegu
  - Konyang University Hospital, Daejeon
  - Namyangju Hanyang General Hospital, Gyeonggi-do
  - Kim Young Ho Internal Medicine Clinic, Gyeongsang
  - Korea University Anam Hospital, Seoul
  - Chung-Ang University Hospital, Seoul